CLINICAL TRIAL: NCT05536999
Title: Follicular FSH Serum Level as a Predictor of an Oocyte Quality and Yield in Fertility Preservation Cycles for Women With a Compromised Ovarian Reserve.
Brief Title: Follicular FSH Serum Level as a Predictor of an Oocyte Yield and Quality in Fertility Preservation Cycles for Women With a Compromised Ovarian Reserve
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Ilana Weizel, Dr Weizel Ilana, Hadassah Medical Organization
Other Study IDs: HMO-0882-22
Record Dates: First submitted 2022-09-08; First posted 2022-09-13 (Actual); Last update posted 2022-10-17 (Actual); Status verified 2022-10

CONDITIONS: Fertility Issues
Keywords: FSH, Social egg freezing, oocyte retrival, follicular fluid , basal FSH, low ovarian reserve
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Blood sample taking , like to measure hormonal level like LH, FSH, Perlakan ,in a follicular fluid after the oocyte retrival — Blood test measure basal FSH, follicular fluid testing

SUMMARY:
The incorporation of ovarian reserve tests in IVF management started after initial publications indicating a potential role for basal FSH in predicting pregnancy outcome after IVF and in counseling patients (1,2). Since these first publications, a large body of additional work on basal FSH and several other tests has been published, often with inconsistent findings on the magnitude and direction of the predictive effect. (3). Level of basal FSH at the start of IVF, in patients aged younger than 40 years, was shown to predict an oocyte yield by several authors, but wasn't related to pregnancy or implantation rates. (4).

Social egg freezing refers to the cryopreservation of mature oocytes on an elective basis for the purpose of delayed childbearing. Many women now have a solution to "bridge the gap between reproductive aging and readiness to have children. Assessment of ovarian reserve enables estimation of the remaining egg pool and can be compared with other women her age. Ovarian reserve tests aim at identifying women at risk of hypo or hyper response to ovarian stimulation: it can possibly detect reproductive lifespan and approximate menopausal timing, assist in counseling family planning and to optimize ovarian response whilst minimizing risks (5).

In Israel, retention of fertility for non-medical reasons is offered for women who have reached the age of 30, but have not yet reached the age of 41. These women may undergo up to 4 retrievals or until 20 eggs are obtained (whichever occurs earlier). The 2022 Health Services, decided to include, for the first-time, to cover cryopreservation for women with a diminished ovarian reserve (6). This unique population is currently addressing our clinic in order to preserve fertility. One of the criteria for coverage entitlement is elevated day 3 FSH level.

The tests used for assessing ovarian reserve include basal day -3 follicle stimulating hormone (FSH, introduced in 1998). Clomiphene citrate challenge test (CCCT, 1989), gonadotropins releasing - hormone agonist stimulation test (GAST, 1989), Inhibin -B (1997), antral follicle count (AFC, 1997) and antimullerian hormone (AMH, 2002.) (7) Measurement of basal FSH is relatively inexpensive, imposes no major burden on the patient, and is widely used in assisted reproductive technology programs.

Follicular fluid provides a very important microenvironment for the development of oocytes. It is reasonable to think that some biochemical characteristics may play a critical role in determining oocyte quality and the subsequent potential to achieve fertilization and embryo development. Components may also provide information on metabolic changes in blood serum, as the circulating biochemical milieu may be reflected in it's composition .

In our current research we wish to assess cycle yield as related to basal FSH level among women diagnosed as having a low ovarian reservoir and were acknowledge as eligible for oocyte cryopreservation coverage. We also would like to measure hormonal level like LH, FSH, Perlakan ,in a follicular fluid after the oocyte retrieval in order to asses the microenvironment .

DETAILED DESCRIPTION:
As a routine monitoring, blood sample is drawn in the early follicular phase (day 3 ). FSH will be documented at this point, prior to IVF cycle initiation. Following this point the treatment will follow routine monitoring including Estradiol measurement, progesteroen measurement and an ultrasound.

Follicular fluid collection: After the laboratory licked the eggs follicular fluid will be aspirated and collected.

The database will include in addition : demographic variables (age, BMI, background morbidities , parity , menstrual parameters ) , number of follicles documented by US ,number of oocytes retrieved number of metaphase II oocytes

Inclusion criteria-

* Ages 30 -41
* Patients who undergo fertility preservation
* Patients with a low ovarian reservoir Exclusion criteria-
* Women with a medical indication for preservation
* Women with a single ovary
* Women planned to undergo in vitro fertilization STATISTICAL ANALYSIS - Descriptive statistics will be used to analyze demographic variables. Correlation coefficients will be used to which evaluate basal FSH , oocyte yield and follicular fluid content . All data will be anonymized prior to data extraction and analysis.

BUDJET- All the laboratory data and ultrasound monitoring are fully covered by the Ministry of Health . Data extraction and analysis will be performed by the IVF unit physicians

ELIGIBILITY:
Inclusion Criteria:

* Fertility preservation patients
* Age 30-41
* Low ovarian reservoir

Exclusion Criteria:

* Women with a single ovary
* Women planned to undergo in vitro fertilization
* Women with cancer diagnosis

Ages: 18 Years to 41 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Women between ages 30 -41, who undergo fertility preservation , were diagnosed as having a low ovarian reservoir and were acknowledge as eligible for oocyte cryopreservation coverage according to the health ministry decision .
Sampling Method: Non-Probability Sample
Enrollment: 64 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Day 3 elevated FSH level is variable in the same patient and is predictive to lower oocyte yield and quality | 2 years
  Measurement of basal FSH in a blood and testing the follicular fluid after oocyte retrieval

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Mount Scoupus, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: Undecided
Every patient receives her own unique number

REFERENCES:
- [Background] Muasher SJ, Oehninger S, Simonetti S, Matta J, Ellis LM, Liu HC, Jones GS, Rosenwaks Z. The value of basal and/or stimulated serum gonadotropin levels in prediction of stimulation response and in vitro fertilization outcome. Fertil Steril. 1988 Aug;50(2):298-307. doi: 10.1016/s0015-0282(16)60077-8. PMID 3135206
- [Background] Roberts JE, Spandorfer S, Fasouliotis SJ, Kashyap S, Rosenwaks Z. Taking a basal follicle-stimulating hormone history is essential before initiating in vitro fertilization. Fertil Steril. 2005 Jan;83(1):37-41. doi: 10.1016/j.fertnstert.2004.06.062. PMID 15652884
- [Background] Bancsi LF, Broekmans FJ, Mol BW, Habbema JD, te Velde ER. Performance of basal follicle-stimulating hormone in the prediction of poor ovarian response and failure to become pregnant after in vitro fertilization: a meta-analysis. Fertil Steril. 2003 May;79(5):1091-100. doi: 10.1016/s0015-0282(03)00078-5. PMID 12738501
- [Background] Al-Azemi M, Killick SR, Duffy S, Pye C, Refaat B, Hill N, Ledger W. Multi-marker assessment of ovarian reserve predicts oocyte yield after ovulation induction. Hum Reprod. 2011 Feb;26(2):414-22. doi: 10.1093/humrep/deq339. Epub 2010 Dec 8. PMID 21147822
- [Background] Revelli A, Delle Piane L, Casano S, Molinari E, Massobrio M, Rinaudo P. Follicular fluid content and oocyte quality: from single biochemical markers to metabolomics. Reprod Biol Endocrinol. 2009 May 4;7:40. doi: 10.1186/1477-7827-7-40. PMID 19413899
- [Background] Behre HM. Clinical Use of FSH in Male Infertility. Front Endocrinol (Lausanne). 2019 May 24;10:322. doi: 10.3389/fendo.2019.00322. eCollection 2019. PMID 31178827
- [Background] Danis RB, Sriprasert I, Ho JR, McGinnis LK, Kumar A, Stanczyk FZ. Association of bioavailable inhibin B and oocyte yield in controlled ovarian stimulation. F S Rep. 2021 Mar 31;2(2):189-194. doi: 10.1016/j.xfre.2021.03.005. eCollection 2021 Jun. PMID 34278353
- [Background] Broer SL, van Disseldorp J, Broeze KA, Dolleman M, Opmeer BC, Bossuyt P, Eijkemans MJ, Mol BW, Broekmans FJ; IMPORT study group. Added value of ovarian reserve testing on patient characteristics in the prediction of ovarian response and ongoing pregnancy: an individual patient data approach. Hum Reprod Update. 2013 Jan-Feb;19(1):26-36. doi: 10.1093/humupd/dms041. Epub 2012 Nov 27. PMID 23188168
- [Background] Leroy JL, Vanholder T, Delanghe JR, Opsomer G, Van Soom A, Bols PE, Dewulf J, de Kruif A. Metabolic changes in follicular fluid of the dominant follicle in high-yielding dairy cows early post partum. Theriogenology. 2004 Sep 15;62(6):1131-43. doi: 10.1016/j.theriogenology.2003.12.017. PMID 15289052
- [Background] Talbot P, Dandekar P. Perivitelline space: does it play a role in blocking polyspermy in mammals? Microsc Res Tech. 2003 Jul 1;61(4):349-57. doi: 10.1002/jemt.10348. PMID 12811740